CLINICAL TRIAL: NCT06283823
Title: Morphological Changes of Removable Orthodontic Retainers During the Use, a Prospective Study
Brief Title: Morphological Changes of Removable Orthodontic Retainers During the Use
Status: Completed | Type: Observational
Sponsor: University of L'Aquila (Other)
Responsible Party: Principal Investigator, Michele Tepedino, Assistant Professor, University of L'Aquila
Other Study IDs: 41821
Record Dates: First submitted 2024-02-21; First posted 2024-02-28 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Orthodontic Retainer
Keywords: orthodontic; retainer; stability; thermoformable retainer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Retainer with high margins: Thermoformed retainers with modified cutout and high margins in the posterior region of the retainer
  Interventions: Device: Thermoformed orthodontic retainer
- Retainer with low margins: Thermoformed retainer with conventional festooned cutout and low margins
  Interventions: Device: Thermoformed orthodontic retainer

INTERVENTIONS:
Device: Thermoformed orthodontic retainer — compare the outcome of the retaining phase of the orthodontic treatment with two different thermoformed retainers

SUMMARY:
The retention is one of the stages of orthodontic treatment that aims to keep the teeth in the correct positions after orthodontic treatment. Without a retention phase, there is a tendency for the teeth to return to their initial position (relapse). To prevent relapse, at the end of orthodontic therapy the use of retaining devices to keep the teeth in their ideal position is required. The aim of the study is to analyse whether intraoral aging of removable retention devices can lead to morphological or dimensional changes, and whether or not these changes are related to orthodontic relapse, expressed as a change in the Peer Assessment Rating (PAR) index. The PAR index is an index that allows us to evaluate the relapse after orthodontic treatment. In this study the PAR index will be measured at the start of the retention period (T0), at the three-months follow-up (T1) and at the six months follow-up (T2). In particular, two types of thermoformed retainers with different cutouts will be evaluated to determine whether the presence of higher margins in a type of retainers allows to maintain greater stability over time and, therefore, to confer a mechanical and clinical advantage.

DETAILED DESCRIPTION:
This study was approved by the Internal Review Board of the University of L'Aquila, L'Aquila, Italy (prot. n. 41821/22). In order to observe a difference between the two groups and the three repeated measurements by ANOVA test equal to a large effect size, with a power of 80% and a probability of the error of the first type equal to 5%, 36 subjects in total will be needed, 18 for each group. Therefore, 36 patients will be selected from the undergraduate students in Dentistry and Oral Hygiene, implementing all the necessary precautions to avoid any problems due to subordination between students participating in the project and teachers.

The eligible patients who will sign a written informed consent, after having received the necessary verbal explanations, will be included in the study. The selected patients will be allocated to one of the two groups (normal masks and masks with modified cutout) by block randomization using Random Allocation Software.

The enrolled patients will be called for the acquisition of a digital impression of the dental arches through an intraoral scanner (CS3600, Carestream Dental LLC, Atlanta, USA). The obtained digital models will be used to create three pairs of identical thermoformed retainers that will be delivered to the patient at a later time. The retainers will be manufactured with custom landmarks at the level of the second molar, between first molar and second premolar, at the level of the canine, and between the two central incisors. Each retainer will be coated with a thin and uniform layer of white paint specially designed to make the material - in itself transparent - scanned with a 5-axis scanner (Zenotec S100, Wieland) obtaining digital copies. Afterwards, the paint will be removed and the retainers will be ready for delivery to the patient.

Patients will be recalled in three steps: T0 (day of delivery of the first retainer), T1 (3 months after delivery) and T2 (9 months after delivery). During the follow-up visits at T1 and T2 new digital scans will be acquired to obtain virtual models of each patient's dental arches. The digital models acquired at T0, T1 and T2 will be used to measure the PAR index according to the Richmond et al. protocol of 1992. This protocol provides for the assignment of a score to the various occlusal parameters that determine a malocclusion, then adding the individual scores to obtain a total score. A score of zero indicates correct alignment and stable occlusion, while positive scores are indicative of a relapse and misalignment.

Patients will be instructed to wear the thermoformed retainers overnight and will receive written instructions on how to clean and manage the retainers, to avoid possible biases due to incorrect procedures. At every subsequent follow-up visits patients will return the used retainers and will receive a new pair. In this way, the first pair of retainers will be used for a total time of three months, while the second pair of retainers will be used for a total time of six months.

To evaluate the morphological changes of the used retainers, their shape and dimensions will be compared to the scanning made before delivery.

After calculating descriptive statistics, the difference between the two retainers type and the three timepoints will be evaluated using a MANCOVA model, after checking for data homoscedasticity with a Levene test.

ELIGIBILITY:
Inclusion Criteria:

* young adult patients: 18-35 years;
* Caucasian ethnic group;
* good oral hygiene (evaluated by observing a plaque index < 20% understood as the sum of the indices of the individual dental elements divided by the number of dental elements considered multiplied by 100);
* patients with normal occlusion Class I occlusion with slight overcrowding and PAR Index less than or equal to 10;
* patients who have received previous orthodontic treatment, with or without stripping;
* patients who have received previous orthodontic treatment with < 20 orthodontic aligners;
* patients who currently use a thermoprinted mask as a restraint, or who do not use any restraint but who would like to receive one.

Exclusion Criteria:

* patients with chromosomal defects, specific neuropsychological disorder, epilepsy (1);
* patients with systemic diseases and comorbidities;
* bruxist patients;
* patients with hypertrophy of chewing muscles, occlusal parafunctions or joint disorders;
* patients with cognitive disabilities with IQ<70;
* patients undergoing drug therapy.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Undergraduate students
Sampling Method: Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2021-12-21 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Peer Assessment Rating (PAR) index | 3 years
  The PAR index will be measured on digital casts to evaluate the amount of alignment relapse.
Volumetric superimposition of digital models | 3 years
  Digital models of pre- and post-usage thermoformed retainers will be superimposed and the distance between the two digital models will be measured

SECONDARY OUTCOMES:
Thickness | 3 years
  The thickness of the material composing the retainers will be measured at different locations.

CONTACTS AND LOCATIONS:
Overall Officials: Michele Tepedino, Principal Investigator — University of L'Aquila
Locations (1):
- University of L'Aquila, L’Aquila, Italy, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Since the data are anonymized it would be acceptable to share it upon reasonable requests.

REFERENCES:
- [Background] Bucci R, Rongo R, Levate C, Michelotti A, Barone S, Razionale AV, D'Anto V. Thickness of orthodontic clear aligners after thermoforming and after 10 days of intraoral exposure: a prospective clinical study. Prog Orthod. 2019 Sep 9;20(1):36. doi: 10.1186/s40510-019-0289-6. PMID 31495908
- [Background] Saghaei M. Random allocation software for parallel group randomized trials. BMC Med Res Methodol. 2004 Nov 9;4:26. doi: 10.1186/1471-2288-4-26. PMID 15535880
- [Background] Schuster S, Eliades G, Zinelis S, Eliades T, Bradley TG. Structural conformation and leaching from in vitro aged and retrieved Invisalign appliances. Am J Orthod Dentofacial Orthop. 2004 Dec;126(6):725-8. doi: 10.1016/j.ajodo.2004.04.021. PMID 15592222
- [Background] Gerard Bradley T, Teske L, Eliades G, Zinelis S, Eliades T. Do the mechanical and chemical properties of InvisalignTM appliances change after use? A retrieval analysis. Eur J Orthod. 2016 Feb;38(1):27-31. doi: 10.1093/ejo/cjv003. Epub 2015 Mar 3. PMID 25740599
- [Background] Lombardo L, Arreghini A, Maccarrone R, Bianchi A, Scalia S, Siciliani G. Optical properties of orthodontic aligners--spectrophotometry analysis of three types before and after aging. Prog Orthod. 2015;16:41. doi: 10.1186/s40510-015-0111-z. Epub 2015 Nov 18. PMID 26582007
- [Background] Thickett E, Power S. A randomized clinical trial of thermoplastic retainer wear. Eur J Orthod. 2010 Feb;32(1):1-5. doi: 10.1093/ejo/cjp061. Epub 2009 Oct 14. PMID 19828592
- [Background] Richmond S, Shaw WC, O'Brien KD, Buchanan IB, Jones R, Stephens CD, Roberts CT, Andrews M. The development of the PAR Index (Peer Assessment Rating): reliability and validity. Eur J Orthod. 1992 Apr;14(2):125-39. doi: 10.1093/ejo/14.2.125. PMID 1582457